CLINICAL TRIAL: NCT05890131
Title: Implementation of Sodium-Glucose Cotransporter (SGLT)-2 Inhibitors in Patients With Heart Failure Through a New Digital Strategy
Brief Title: Implementation of SGLT-2 Inhibitors in Patients With Heart Failure Through a New Digital Strategy
Acronym: EMAIL-HF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Morten Schou (Other)
Responsible Party: Sponsor-Investigator, Morten Schou, MD, PhD, Professor, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: P-2022-675
Record Dates: First submitted 2023-05-03; First posted 2023-06-06 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure
Keywords: Heart Failure; SGLT-2 inhibitors; Digital implementation; Cardiorenal disease
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the trial design, blinding the patients who received the digital letters is not possible. However, the letters do not disclose that they were sent as part of a randomized trial, which enhances the generalizability of the study intervention. Additionally, patients in the control group, who did not receive a letter, remain unaware that they are part of the control group in a randomized trial. Also, the HF specialists who prescribed the SGLT2 inhibitors are blinded to the primary endpoint, as they do not receive information on whether patients actually redeemed their prescriptions and commenced the medication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital letter (Experimental): The experimental group will receive a digital letter with information on the newly approved heart failure therapy option, SGLT-2 inhibitors. The letter will also invite recipients to be evaluated by a heart failure specialist for potential initiation of the therapy.
  Interventions: Other: Digital letter
- Control (No Intervention): The control group will not be sent the digital letter and will therefore receive usual follow-up and care in the public healthcare system.

INTERVENTIONS:
Other: Digital letter — A digital letter with evidence-based information about the newly approved heart failure therapy option, SGLT-2 inhibitors. The letter will also invite recipients to be evaluated by a heart failure specialist for potential initiation of the therapy.
  Arms: Digital letter

SUMMARY:
The implementation of new medical therapies and guidelines, is a long and complex process that takes up to 10 years on average. This prolonged process is a global challenge and is mainly due to the complexity of cross-institutional patient care, involving primary care, out-patient clinics, nursing homes and patient associations.

The main objective of this clinical trial is to determine whether a new digital strategy that employs official digital letters to inform and invite patients to evaluate their eligibility for new therapies, specifically the sodium-glucose co-transporter-2 (SGLT-2) inhibitor for heart failure patients, can facilitate and optimise the implementation. The aim is to increase the number of eligible patients with heart failure who start taking SGLT-2 inhibitors and reduce the time it takes to initiate treatment compared to the current process. Ultimately, this approach may improve patient outcomes.

DETAILED DESCRIPTION:
The study is a prospective, multicenter, two-armed, randomised clinical trial that will be coordinated from the Department of Cardiology, Herlev-Gentofte Hospital. The primary objective of the study is to determine whether a new digital strategy can be implemented to introduce novel medical therapies, specifically sodium-glucose co-transporter-2 (SGLT-2) inhibitors to heart failure patients. The aim is to increase the number of eligible patients who initiate therapy and to reduce the time taken to initiate therapy compared to the current process. The study will recruit patients with a registered diagnosis of heart failure residing in The Capital Region of Denmark and Roskilde, who have not yet been started on SGLT-2 inhibitor therapy. Patient identification and recruitment will be carried out through Danish nationwide registries, using their personal identification number (CPR-number), which is also linked to a secure digital mailbox where all official letters from public authorities are sent to Danish citizens. Patients will be randomly assigned (1:1) to receive a digital letter containing evidence-based information about the newly approved heart failure therapy option, SGLT-2 inhibitors. The letter will also invite recipients to be evaluated by a heart failure specialist for potential initiation of the therapy. Outcome measures will be obtained from Danish nationwide registers at pre-specified time points and in collaboration with the Danish Health Data Authority.

ELIGIBILITY:
Inclusion Criteria:

1. Registered diagnosis of heart failure within the last 10 years
2. Living in the Capital Region of Denmark or Roskilde
3. Age ≥20 years

Exclusion Criteria:

1. Redeemed prescription of a SGLT-2 inhibitor after 2015
2. Type 1 diabetes
3. History of diabetic ketoacidosis
4. Chronic kidney disease in long term dialysis
5. Living in a nursing home
6. Dementia
7. Cancer diagnosis within the last year (except prostate cancer and non-melanoma skin cancer)
8. Exemption from the public digital mailbox system

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5996 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients initiating therapy with a SGLT-2 inhibitor | from randomisation up to 6 months

SECONDARY OUTCOMES:
Time to first occurrence of a composite heart failure endpoint consisting of all-cause death or heart failure hospitalisation. | from randomisation up to 2 years

OTHER OUTCOMES:
Number of all-cause deaths and heart failure hospitalisations | from randomisation up to 2 years
Time to first occurrence of a 3-point expanded composite heart failure endpoint consisting of all-cause death, heart failure hospitalisation, or renal failure, with examination of the components of this composite. | from randomisation up to 2 years
Time to first occurrence of a 4-point expanded composite heart failure endpoint consisting of all-cause death, heart failure hospitalisation, non-fatal myocardial infarction, non-fatal stroke, with examination of the components of this composite. | from randomisation up to 2 years
Time to initiation of SGLT-2 inhibitor therapy | from randomisation up to 2 years
Adherence to SGLT-2 inhibitor therapy (defined as proportion of days covered >=80%) | from randomisation up to 1 year
Proportion of elderly (>75 years) initiating therapy with SGLT-2 inhibitors | from randomisation up to 2 years
Proportion of patients with lower educational level initiating therapy with SGLT-2 inhibitors | from randomisation up to 2 years
Proportion of patients with lower socioeconomic level initiating therapy with SGLT-2 inhibitors | from randomisation up to 2 years
Proportion of immigrants initiating therapy with SGLT-2 inhibitors | from randomisation up to 2 years
Proportion of patients with type 2 diabetes initiating therapy with SGLT-2 inhibitors | from randomisation up to 2 years
Proportion of male and female patients initiating therapy with SGLT-2 inhibitors | from randomisation up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Morten Schou, MD, PhD, Principal Investigator — Department of Cardiology, Herlev and Gentofte Hospital, 2900 Hellerup, Denmark; Lars Køber, MD, DMSc, Study Chair — Department of Cardiology, Rigshospitalet, Blegdamsvej 9, 2100 Copenhagen, Denmark
Locations (5):
- Denmark (5):
  - Bispebjerg-Frederiksberg Hospital, Copenhagen
  - Herlev and Gentofte University Hospital, Hellerup
  - Nordsjællands Hospital, Hillerød
  - Amager-Hvidovre-Glostrup Hospital, Hvidovre
  - Sjællands Universitetshospital - Roskilde, Roskilde

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected from nationwide administrative registers, that are stored and managed by the Danish Health Data Authority. Data access can only be made available to a third party through an affiliation to an authorized Danish research environment. Please contact the sponsor-investigator in case of any inquiries.